CLINICAL TRIAL: NCT04752787
Title: The Effect of QR Code Supported Online Breastfeeding Training Given to Pregnant Women Expecting Twin Babies on Breastfeeding Intention and Feeding With Breast Milk in the First Six Months
Brief Title: Effect of Breastfeeding Training
Acronym: Breastfeeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, dilek menekşe, Assistant professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Dilek MENEKŞE
Record Dates: First submitted 2021-01-26; First posted 2021-02-12 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Breastfeeding
Keywords: Twin Baby; Twin Pregnancy; Quick Response Code; Breastfeeding Training; Breastfeeding Intention
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Since the education about twin babies breastfeeding will be given by the researchers, single-blind randomization will be provided.
  The statistician will also be made blind for the data analysis purpose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental (Experimental): Experimental group 1: Breastfeeding training for successful breastfeeding in twin babies will be given to the online training group. The training will be carried out by the researchers (DM) and (SYC) using visual training tools (power point presentation, simultaneous breastfeeding animations in twin babies and breastfeeding guide). Due to the Covid-19 pandemic process, it will be carried out online and remotely. Training on successful breastfeeding in twin babies will be carried out in two sessions at a time. In the first session, about 45 minutes of online slide-assisted training on successful breastfeeding in twin babies and the importance of breast milk will be conducted and questions of pregnant women will be answered. Total training will take approximately one and a half hours.
  Interventions: Other: Online breastfeeding training
- Active comparator (Active Comparator): Experimental group 2: Breastfeeding training for successful breastfeeding in twin babies will be given to the QR supported online training group. Due to the Covid-19 pandemic process, it will be carried out online and remotely. Training on successful breastfeeding in twin babies will be carried out in two sessions at a time. Total training will take approximately one and a half hours.
  In the guideline, there will be 4 vieos ralted to "Breastfeeding and Feeding with Breast Milk in Twin Babies", "Breastfeeding Techniques and Positions in Twin Babies", "Expressing Breastfeeding, Storing and Feeding it to Babies" and "Problems Encountered in Breastfeeding and its Solutions", and simultaneous breastfeeding used in breastfeeding twin babies and also there will be a total of 7 QR codes, 3 of which are related to the animations (Animation 1-2-3) of the positions (double cradle grip, double football grip, combination of armpit and cradle grip-parallel grip).
  Interventions: Other: QR code supported online breastfeeding training
- Control Groups (No Intervention): Pregnant women in the control group will be followed up in line with the routine health monitoring and information of the hospital.

INTERVENTIONS:
Other: Online breastfeeding training — Online breastfeeding training will be provided to pregnant women expecting twin babies.
  Arms: Experimental
Other: QR code supported online breastfeeding training — QR code supported online breastfeeding training will be given to pregnant women who are expecting twin babies.
  Arms: Active comparator

SUMMARY:
Breast milk is a unique, natural and universal food with excellent content that ensures healthy growth and development of the baby. Since twin babies are mostly born prematurely, with low birth weight and with health problems affecting important systems such as respiratory and gastrointestinal systems, breastfeeding becomes more important. Studies show that mothers with twin babies can produce sufficient quantity and quality of milk. However, the breastfeeding rates of twin babies are not at the desired level. In the successful breastfeeding of twin babies, breastfeeding education started before birth has an important place in initiating and maintaining successful breastfeeding. Today, it is recommended to use different materials and techniques in order to ensure continuity in the training given to healthy and sick individuals. One of them is QR code supported training. Using different training and method techniques will make it easier for nurses to be more effective. The aim of this study is to examine the effect of QR code supported online breastfeeding education given to pregnant women expecting twins on breastfeeding intention and feeding with breast milk in the first six months.

Research Hypotheses:

H0: There is no difference between breastfeeding intention and success of mothers who have twin babies who are given online breastfeeding training and those who are not.

H1: The breastfeeding intention and success of mothers with twin babies who are given online breastfeeding training with QR code is higher than mothers who are given online breastfeeding training only.

H1: The breastfeeding intention and success of mothers with twin babies who are given online breastfeeding training with QR code is higher than mothers who are not given breastfeeding training.

DETAILED DESCRIPTION:
Background: With the increase in the use of assisted reproductive techniques thanks to the studies and developing technology in recent years, a significant increase has been observed in multiple pregnancy rates. Studies conducted in the world and in our country have stated that the twin birth rate is between 1.86-10.9%. With the increase in twin pregnancies evaluated in the risky pregnancy group, the responsibilities of healthcare professionals on issues such as regular follow-up in both antenatal and postnatal periods, ensuring successful breastfeeding, and care of babies have increased.

Breast milk is the most appropriate and valuable food source for multiple babies like single babies. Although there is strong evidence about the benefits of breast milk, it has been emphasized in studies that the rate and duration of breastfeeding in twin babies are low and not at the desired level compared to single babies. Although there are many factors affecting these rates, the most important one is the mother's decision and intention to breastfeed her babies during pregnancy. During the mother's pregnancy; The feeling of uncertainty and inadequacy about birth, feeding and care of the baby causes loss of trust in the mother and results in unwanted experiences by affecting her motivation.This situation can be further complicated by the thought of being a twin mother. Therefore, the continuation of breastfeeding training that started before birth in the postnatal period in line with the needs of the mothers, and individualized breastfeeding support have an important role in the initiation and maintenance of successful breastfeeding.

Today, it is recommended to use different materials and techniques in order to ensure continuity in the training given to healthy and sick individuals. One of them is QR code supported training. Quick Response (QR) codes, which act as a bridge between old and new educational materials, make the learning process more permanent with visual materials by providing instant access to different media applications such as audio, image and video, beyond reading texts and reading the resources at any time. For this reason, QR Codes increase the effectiveness of the training by giving booklets during the education of expectant mothers, as well as satisfying the participants who are interested in traditional learning methods, while at the same time increasing the effectiveness of the learned theoretical knowledge to be practiced by following it practically at the desired time and place. QR codes also for organizations in developing countries such as Turkey have limited resources available can be integrated easily because it requires high cost and user-provided printed materials instantly accessible. QR codes, which are integrated into the booklet used in neonatal care education, because they require theory and skills, facilitate access to videos and enable the acquisition and adoption of many care practices with the interaction of image, sound and movement supported by mobile applications. In addition, considering the rapid increase in the use of smart phones today, mobile applications have a significant effect in improving health in order to increase the quality of health services. The cost-effectiveness of mobile applications, enabling individuals to learn whenever they want and appropriate for themselves without limitation of time and space, allowing individuals to follow-up and training at any time and being accessible make these applications more attractive.

In this extraordinary period in which we have experienced the COVID-19 pandemic, which has deeply affected the world recently, the need to review health education methods, especially for vulnerable groups such as pregnant women, has arisen due to the risk of hospital environments. This method we offer will be effective in ensuring safe health education and continuity. The QR Code application can also be used by integrating into different healthy / sick individual trainings, thus reducing the workload of healthcare professionals.

In the light of this information; The study was planned to determine the effect of QR code supported online breastfeeding training given to pregnant women expecting twins on breastfeeding intention and feeding with breast milk in the first six months.

Method: This research is a randomized controlled experimental study. The sample of the study will be visited between the dates of 01.02.2021-01.02.2022 to the pregnant outpatient clinics of the Sakarya Maternity and Children's Hospital Campus of the Ministry of Health Sakarya University Training and Research Hospital. It will create twin pregnancies between the week of gestation. Power analysis was performed using the G * Power (v3.1.7) program to determine the sample size. When it is not known how many units of difference between groups are important, the effect width value is taken as 0.70 as the method used. The effect width value is 0.20 very high, 0.50 medium level, and 0.80 gives the results under the maximum acceptance constraint. It means that the higher the power of the study, the more precise the measurement is in finding the difference. Power is expected to be 0.80 and above. However, some experts emphasize that this limit is between 0.70 and 0.90. The study was planned with a total of 102 pregnant women, 34 babies for each group, when the probability of type 1 error (α) was 0.05 (95% confidence level), 80% power level and the effect width value was 0.70. A total of 102 pregnant women that make up the sample in the study will be randomly divided into three groups. Pregnant women to be assigned to the groups will be assigned through a computer-based random number generator program.

The sample of the study will randomly allocated into three groups: online training for intervention group-1, online training with QR code support for intervention group-2 and the other group, which was the control group, routine health monitoring of the hospital and will be followed in line with their information. Since the education about twin babies breastfeeding will be given by the researchers, single-blind randomization will be provided. The statistician also will be made blind for the data analysis purpose. In data collection tools, "Descriptive Information Form" containing sociodemographic characteristics of the family, "Breastfeeding Intention Scale in Pregnant Women Expecting Twin Babies" to measure the breastfeeding intention of pregnant women who are expecting twin babies, and the babies created by researchers to monitor breastfeeding status in the postnatal period. will be collected using the "Breastfeeding Follow-up Chart", which includes birth histories, hospital stays and breastfeeding processes.

The first stage of the study includes the training and filling out the "Introductory Information Form" and the Breastfeeding Intention Scale for Pregnant Women Expecting Twin Babies "before the training. The training to be given to the experimental groups (intervention 1: Online training group, intervention - 2: Online training group with QR code support) will be carried out online and remotely. Training on successful breastfeeding in twin babies will be carried out in two sessions at a time. Powerpoint presentation, simultaneous breastfeeding animations for twin babies, breastfeeding guide will be used as educational materials. In addition, QR codes will be integrated into the guide in order to provide the opportunity to watch the video simultaneously while reading the guide in situations that require knowledge and skills related to breastfeeding and to allowed them to watch repeatedly as long as they feel the need. QR Codes for Videos on Breastfeeding Training in Twin Pregnants will only be used in the intervention - 2: QR supported Online training group. The training will take approximately 1.5 hours on average. After the training, the questions of the pregnant women will be answered. Before the pregnant women leave the training, breastfeeding guide will be sent to the intervention 1 group, and the training guide with QR code to the intervention 2 group will be sent to the e-mails of the pregnant women. The pregnant women in the Intervention 2 group will be periodically sent reminder notifications to watch the videos before and after the birth via the QR Codes in the guide. No intervention will be made to the control group. The second phase of the study includes the postnatal breastfeeding follow-up of pregnant women. At this stage, the pregnant women will be called every month starting from the 1st month to the 6th month in the first week after giving birth, and the nutritional status of the babies in the first 6 months will be followed by using the "Breastfeeding Follow-up Chart" form. In the evaluation of data, statistical analysis will be performed using the SPSS package program. The Kolmogorov-Smirnov (K-S) test will be used for normality. In order to determine whether there is a difference in the dependent variables compared to independent variables, the independent group t-test will be used if the distribution is normal in independent variables with two options, and Mann Whitney-U test will be used if distribution is not normal. The results will be evaluated at a confidence level of 95% and at a level of significance of p <0.05.

ELIGIBILITY:
Inclusion Criteria:

Twin pregnant women who come to the pregnancy outpatient clinic

* Having twin babies after birth,
* Whose are least literate,
* Pregnant women who can speak and understand Turkish well
* Whose are 19 years of age or older,
* Volunteering to participate in research,
* Whose are between 28 -34th weeks of gestation,
* Whose been Primigravida and her pregnancy twin
* Do not have a diagnosed neurological, psychiatric or chronic disease (diabetes, chronic kidney failure, etc.) that will affect breastfeeding.
* No health problems in mother and babies before or after birth
* Risky drug use that passes through breast milk after birth
* Pregnant women who have a smart phone, computer, tablet and wireless internet will be included in the study.

Exclusion Criteria:

Whose are 18 years of age or under Whose been multigravida and / or multiparous Whose have any health problems in the mother and babies before or after birth Whose do not have a smart phone, computer, tablet or wireless internet during the study period Participants who complete the questionnaire forms as missing will be excluded from the study.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — mothers
Enrollment: 102 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of breastfeeding intention in study and control groups | Change from pre-education and two weeks after education breastfeeding intention
  Breastfeeding Intention Scale for Pregnant Expecting Twin Babies" developed to evaluate the intention of breastfeeding in pregnant women expecting twin babies, each item is scored from 1 to 5 on a 5-point Likert-type scale consisting of 7 positive items and the scores vary according to the responses of the items. Scoring items; Strongly Disagree (1), Disagree (2), Moderately Agree (3), Agree (4), Strongly Agree (5). The minimum score that can be obtained from the scale is 7 and the maximum score is 35. The high total score obtained from the scale indicates that pregnant women expecting twin babies have a high breastfeeding intention.

SECONDARY OUTCOMES:
Breastfeeding rates in study and control groups | Within the first week following the birth of pregnant women, every month starting from the 1st month until the 6th month
  Proportion who report giving any breastmilk within the past 24 hours
Exclusively breastfeeding rates in study and control groups | Within the first week following the birth of pregnant women, every month starting from the 1st month until the 6th month
  Proportion who report only giving breastmilk within the past 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Menekşe, Ass.prof., Study Director — Sakarya University; Sinem Yalnızoğlu Çaka, Res. Asist. Dr., Principal Investigator — Sakarya University; Nursan Çınar, Prof. Dr., Principal Investigator — Sakarya University; Hilal Uslu Yuvacı, Assist. prof., Principal Investigator — Sakarya University; Bilge Kapudere, Res. Asist. Dr., Principal Investigator — Sakarya University
Locations (1):
- Sakarya University, Sakarya, Serdivan, Turkey (Türkiye)

REFERENCES:
- [Background] Güler, E., & Eby, G. (2015). Akıllı ekranlarda mobil sağlık uygulamaları. Eğitim ve Öğretim Araştırmaları Dergisi, 4(3), 45-51.
- [Background] Al Saleh, S., & Bhat, S. A. (2015). Mobile learning: A systematic review. International Journal of Computer Applications, 114(11), 1-5.
- [Background] Samples, C., Ni, Z., & Shaw, R. J. (2014). Nursing and mHealth. International Journal of Nursing Sciences, 1(4), 330-333. https://doi.org/10.1016/j.ijnss.2014.08.002
- [Background] Aktaş, C., & Çaycı, B. (2013). QR kodun mobil eğitimde yeni eğitim yöntemlerinin geliştirilmesine katkısı. Global Media Journal, 119, 1-5.
- [Background] Hau, G. B., Siraj, S., Alias, N., Rauf, R. A. A., & Zakaria, A. (2013). Research and trends in the field of technology-enhanced learning from 2006 to 2011: A content analysis of Quick Response Code (QR-Code) and ıts application in selected studies. Malaysian Online Journal of Educational Technology, 1(1), 54-72. Retrieved from https://files.eric.ed.gov/fulltext/EJ1086361.pdf
- [Background] Overdijkink SB, Velu AV, Rosman AN, van Beukering MD, Kok M, Steegers-Theunissen RP. The Usability and Effectiveness of Mobile Health Technology-Based Lifestyle and Medical Intervention Apps Supporting Health Care During Pregnancy: Systematic Review. JMIR Mhealth Uhealth. 2018 Apr 24;6(4):e109. doi: 10.2196/mhealth.8834. PMID 29691216
- [Background] Yayla M, Baytur Y. (2008). Multicentric multiple pregnancy study I - Epidemiology. Prenatal Journal, 16 (1): 1-8.
- [Background] Türkiye Neonataloji Derneği Yardımlı Üreme Teknikleri ve Çoğul Gebelikler Çalışma Grubu (2010). Yardımlı Üreme tekniklerinin neonatal mortalite ve morbidite üzerine etkileri. Çocuk Sağlığı ve Hastalıkları Dergisi, 53: 258-266.
- [Background] Sezer SD, Kucuk M, Yuksel H, Odabasi AR, Turkmen M, Cakmak BC, Doger FK. Perinatal and neonatal outcomes of twin pregnancies in Turkey. Twin Res Hum Genet. 2011 Apr;14(2):201-12. doi: 10.1375/twin.14.2.201. PMID 21425905
- [Background] Martin JA, Hamilton BE, Osterman MJ, Driscoll AK, Mathews TJ. Births: Final Data for 2015. Natl Vital Stat Rep. 2017 Jan;66(1):1. PMID 28135188
- [Background] Saint L, Maggiore P, Hartmann PE. Yield and nutrient content of milk in eight women breast-feeding twins and one woman breast-feeding triplets. Br J Nutr. 1986 Jul;56(1):49-58. doi: 10.1079/bjn19860084. PMID 3676208
- [Background] Ooki S. Breast-feeding rates and related maternal and infants' obstetric factors in Japanese twins. Environ Health Prev Med. 2008 Jul;13(4):187-97. doi: 10.1007/s12199-008-0028-y. Epub 2008 Apr 22. PMID 19568905
- [Background] Ostlund A, Nordstrom M, Dykes F, Flacking R. Breastfeeding in preterm and term twins--maternal factors associated with early cessation: a population-based study. J Hum Lact. 2010 Aug;26(3):235-41; quiz 327-9. doi: 10.1177/0890334409359627. Epub 2010 Feb 5. PMID 20139377
- [Background] Whitford HM, Wallis SK, Dowswell T, West HM, Renfrew MJ. Breastfeeding education and support for women with twins or higher order multiples. Cochrane Database Syst Rev. 2017 Feb 28;2(2):CD012003. doi: 10.1002/14651858.CD012003.pub2. PMID 28244065
- [Background] Basu S, Aundhakar CD, Galgali A. (2014). Gender discrimination in relation to exclusive breast feeding practices amongst twins in Rural India. International Journal of Health Sciences & Research, 4 (5): 139-43.
- [Background] Cinar N, Kose D, Alvur M, Dogu O. Mothers' Attitudes Toward Feeding Twin Babies in the First Six Months of Life: A Sample From Sakarya, Turkey. Iran J Pediatr. 2016 Jun 14;26(5):e5413. doi: 10.5812/ijp.5413. eCollection 2016 Oct. PMID 28203331
- [Background] Damato EG, Dowling DA, Madigan EA, Thanattherakul C. Duration of breastfeeding for mothers of twins. J Obstet Gynecol Neonatal Nurs. 2005 Mar-Apr;34(2):201-9. doi: 10.1177/0884217504273671. PMID 15781597
- [Background] Bennington LK. (2011). Breastfeeding multiples: It can be done. Newborn Infant Nurs Rev, 11: 194-197.
- [Background] Langkamp DL, Girardet RG. Primary care for twins and higher order multiples. Curr Probl Pediatr Adolesc Health Care. 2006 Feb;36(2):47-67. doi: 10.1016/j.cppeds.2005.10.005. No abstract available. PMID 16414559
- [Background] Odei AB. (2013). Factors Assocıated with Exclusive Breastfeeding of Ghanaian Twins. The Unıversity of Ghana, Ghana, (Principal Supervisor: Prof Anna Lartey, Co-Supervisor: Dr. Gloria Ethel Otoo)
- [Background] Yenal K, Tokat MA, Ozan YD, Çeçe Ö, Abalın FB. (2013). Annelerin emzirme öz-yeterlilik algıları ile emzirme başarıları arasındaki ilişkinin incelenmesi. Hemşirelikte Eğitim ve Araştırma Dergisi, 10 (2): 14-19.
- [Background] Lumbiganon P, Martis R, Laopaiboon M, Festin MR, Ho JJ, Hakimi M. Antenatal breastfeeding education for increasing breastfeeding duration. Cochrane Database Syst Rev. 2016 Dec 6;12(12):CD006425. doi: 10.1002/14651858.CD006425.pub4. PMID 27922724
- [Background] Shim JI, Kang SJ. Impact of Breastfeeding Knowledge, Attitude, and Barriers on Breastfeeding Practice among Twin Mothers. Korean J Women Health Nurs. 2017 Jun;23(2):89-98. doi: 10.4069/kjwhn.2017.23.2.89. Epub 2017 Jun 27. PMID 37684888
- Available data/document: Study Protocol — http://files.eric.ed.gov/fulltext/EJ1086361.pdf
- Available data/document: Study Protocol — https://mhealth.jmir.org/2018/4/e109/